CLINICAL TRIAL: NCT05976451
Title: Time Effect on the Predictability of Different Grafting Materials in Treatment of Gingival Recession RT 1in the Esthetic Zone
Brief Title: Time Effect on the Predictability of Different Grafting for Gingival Recession RT 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mahetab mohamed abdel el wahab, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1011
Record Dates: First submitted 2023-03-12; First posted 2023-08-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-07

CONDITIONS: Gingival Recession Types One(RT1)
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- collagen matrix (Experimental): melatonin in collagen matrix with Modified Coronally Advanced Tunneling Technique (MCAT)
  Interventions: Combination Product: melatonin with collagen matrix
- connective tissue graft (CTG) (Active Comparator): connective tissue graft with Modified Coronally Advanced Tunneling Technique (MCAT)
  Interventions: Combination Product: connective tissue graft (CTG)

INTERVENTIONS:
Combination Product: melatonin with collagen matrix — (CMX) with melatonin in the esthetic zone using Modified Coronally Advanced Tunneling Technique (MCAT)
  Arms: collagen matrix
Combination Product: connective tissue graft (CTG) — control group connective tissue graft using Modified Coronally Advanced Tunneling Technique (MCAT)
  Arms: connective tissue graft (CTG)

SUMMARY:
The primary objective of this study was to evaluate time effect on the clinical predictability of collagen matrix Xenograft (CMX) with melatonin gel versus connective tissue graft (CTG) and determine whether it is proposed to be an alternative in multiple adjacent gingival recession (MAGR) in recession type one (RT1)

DETAILED DESCRIPTION:
this study was conducted to evaluate time effect on the clinical predictability of collagen matrix Xenograft (CMX) with melatonin gel versus connective tissue graft (CTG) and determine whether it is proposed to be an alternative in multiple adjacent gingival recession

ELIGIBILITY:
Inclusion Criteria:

* Presence of RT1 GRs of the maxillary or mandibular arch in the esthetic zone with a GR depth ≥2 mm,
* patients >18 years old,
* Full mouth plaque index score <20%
* Systemically and periodontally healthy patients.

Exclusion Criteria:

* Smokers
* Patients with periodontitis stage III and IV were previous surgical treatment of GR,
* Pregnant or breastfeeding women; P
* Patients with para-functional habits or any source of occlusal trauma.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
interproximal clinical attachment level | 6-9 months
  measured from CEJ to base of pocket depth by using periodontal prob
Probing pocket depth (PPD) | 6-9 months
  from gingival margin to pocket depth measured by mm
Recession depth | 6-9 months
  measure from CEJ to gingival margin by mm

SECONDARY OUTCOMES:
Keratinized tissue width | 6-9 months
  from free gingival groove to MGJ

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt